CLINICAL TRIAL: NCT06877390
Title: Effect of Enhanced External Counterpulsation on the Rehabilitation of Patients With Acute Myocardial Infarction After Drug-Coated Balloon-Based Percutaneous Coronary Intervention
Brief Title: Effect of Enhanced External Counterpulsation
Acronym: EECP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongming Hospital Affiliated to Shanghai University of Health & Medicine Sciences (Other)
Responsible Party: Principal Investigator, Yingmin Lu, Principal Investigator, Chongming Hospital Affiliated to Shanghai University of Health & Medicine Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ChongmingHospital
Record Dates: First submitted 2025-02-12; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Enhanced External Counterpulsation (EECP); Acute Myocardial Infarction (AMI); Drug-coated Balloon; Cardiac Rehabilitation
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): During the observation period after undergoing DCB-based PCI, patients in the control group received antiplatelet agents (100 mg of aspirin and 75 mg of clopidogrel, once a day), β-blocker (25-100 mg of metoprolol, twice a day, with the dose adjusted based on the patient's heart rate) and statins (10-20 mg of rosuvastatin, every night). In addition, the patients received exercise rehabilitation (e.g. aerobic, resistance and flexibility training) for 30-60 min, 3-5 times/week.
  Interventions: Other: conventional drug and exercise rehabilitation
- Rehabilitation group (Experimental): Patients in the rehabilitation group received the same medication and exercise rehabilitation as the control group during the trial period after undergoing DCB-based PCI DCBs; in addition, they were provided with EECP treatment after 7 days of medication. The treatment adopted a P-ECP/TI EECP device with a pressure setting of 0.020-0.035 MPa. Based on patients' actual tolerance, the treatment pressure and inflation and exhaust times were adjusted to a diastolic/systolic blood pressure ratio of >1.2 and a diastolic/systolic pressure area of 1.5-2.0. The treatment was applied daily for 1 hour, 6 days a week, for a total of 36 hours.
  Interventions: Device: EECP-based rehabilitation regimen

INTERVENTIONS:
Other: conventional drug and exercise rehabilitation — patients in the control group received antiplatelet agents (100 mg of aspirin and 75 mg of clopidogrel, once a day), β-blocker (25-100 mg of metoprolol, twice a day, with the dose adjusted based on the patient's heart rate) and statins (10-20 mg of rosuvastatin, every night). In addition, the patients received exercise rehabilitation (e.g. aerobic, resistance and flexibility training) for 30-60 min, 3-5 times/week.
  Arms: Control group
Device: EECP-based rehabilitation regimen — Patients in the rehabilitation group received the same medication and exercise rehabilitation as the control group during the trial period after undergoing DCB-based PCI DCBs; in addition, they were provided with EECP treatment after 7 days of medication. The treatment adopted a P-ECP/TI EECP device with a pressure setting of 0.020-0.035 MPa. Based on patients' actual tolerance, the treatment pressure and inflation and exhaust times were adjusted to a diastolic/systolic blood pressure ratio of >1.2 and a diastolic/systolic pressure area of 1.5-2.0. The treatment was applied daily for 1 hour, 6 days a week, for a total of 36 hours.
  Arms: Rehabilitation group

SUMMARY:
This study evaluated the efficacy and safety of enhanced extracorporeal counterpulsation for cardiac rehabilitation in patients after DCB for acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* patients with AMI diagnosed based on the universal definition of myocardial infarction criteria
* a single vessel infarcted, and Syntax score ≤22
* patients treated using DCB
* patients without EECP contraindications
* patients aged 18-75 years
* patients who had signed informed consent and were able to cooperate in completing the study

Exclusion Criteria:

* patients with lower limb deep venous thrombosis and active thrombophlebitis
* patients with moderate to severe valvular heart disease, especially those with aortic insufficiency and/or stenosis
* patients with moderate to severe pulmonary arterial hypertension (mean pulmonary arterial pressure >50 mmHg)
* patients with aortic, cerebral or dissecting aneurysms
* patients with uncontrolled hypertension (>180/110 mmHg)
* patients with decompensated heart failure (cardiac function of grade IV)
* patients with arrhythmia that might interfere with the electrocardiographic gating function of the EECP device
* patients with haemorrhagic diseases or obvious bleeding tendencies
* patients with infected lesions in their limbs that may affect EECP
* pregnant women
* patients with ventricular aneurysm and mural thrombus detected through echocardiography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of baseline data | followed up for 6 months
  Patients' gender
Comparison of baseline data | followed up for 6 months
  Patients' age
Comparison of baseline data | followed up for 6 months
  Patients' body mass index
Comparison of baseline data | followed up for 6 months
  Patients' smoking and drinking history
Comparison of baseline data | followed up for 6 months
  Patients' comorbidities (hypertension, diabetes and hyperlipidaemia)
Comparison of baseline data | followed up for 6 months
  Patients' infarcted vessels
Comparison of baseline data | followed up for 6 months
  Patients' preoperative NYHA cardiac function grading
Comparison of baseline data | followed up for 6 months
  Patients' CCS angina grading
Comparison of cardiac function | followed up for 6 months
  In the indicators, including the CO, SV and LVEF
Comparison of brain natriuretic peptide levels | followed up for 6 months
  BNP levels.
Comparison of 6-minute walking distance | followed up for 6 months
  The 6MWD in the rehabilitation group.
Comparison of cardiac function gradings | followed up for 6 months
  The New York Heart Association（NYHA ）scale classifies impaired heart function into four levels according to the degree of activity that triggers symptoms of heart failure. A higher grade indicates more severe symptoms.
Comparison of cardiac angina gradings | followed up for 6 months
  The Canadian Cardiovascular Society (CCS) grading system for angina pectoris is divided into four levels, with different treatment options. A higher grade indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- P-ECP/TI EECP device, Shanghai, China

IPD SHARING:
Plan to Share IPD: No